CLINICAL TRIAL: NCT05737238
Title: Evaluation of a Compensatory Brain Game Supporting Goal Management Training Targeting Executive Function After Acquired Brain Injury Using Single-case Experimental Design Methodology
Brief Title: A Single-case Design to Investigate a Compensatory Strategy Game Supporting Goal Management Training
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Klimmendaal Revalidatiespecialisten (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Karman Line GMT SCED
Record Dates: First submitted 2022-12-02; First posted 2023-02-21 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-02

CONDITIONS: Acquired Brain Injury; Executive Dysfunction; Goal Management Training; Compensatory Strategy Training; Serious Gaming
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Intervention Model Description: A randomized Single-case Experimental Design (SCED) with a follow-up period of 1 month. Participants will be first assigned to a baseline phase (phase A). The start of the treatment phase (phase B) is determined randomly for each participant, given the restriction that the baseline phase (phase A) should last for at least three weeks (21 days) and at most five weeks (30 days). This means that the treatment phase can start on any day between the 21th and the 30th days. So, in the first three weeks, all participants are in the baseline condition. The duration of baseline will thus be different for each subject. Nonspecific effects, such as linear trends, retesting or non-specific recovery, can be controlled by this approach, since expected changes in level of performance due to treatment should parallel this stepwise onset of therapy procedure.
  Phase A acts as a control and is therefore compared with phase B.
Who Masked: Outcomes Assessor
Masking Description: The target behavior (i.e. performance on an untrained shopping task) will be measured repeatedly, on a minimum of six occasions in each phase where possible, in accordance with the recommendations of the What Works Clearinghouse and RoBiNT criteria (Tate et al., 2013). Repeated measures of target behavior will be assessed via the OxMET-NL task and is scored automatically: no assessor input is required to either save or score the main outcome data. The secondary outcome measure(s) are scored by an outcome assessor who is blind to the order in which the secondary outcome measure(s) were taken.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Baseline phase (Phase A) (No Intervention): At the start of the study, all participants are assigned to the baseline phase (phase A). During phase A, patients do not receive interventions related to executive function problems. The start of the intervention phase (phase B) is determined randomly for each participant, given the restriction that phase A should last for at least three weeks (21 days) and at most five weeks (30 days). This means that phase B can start on any day between the 21th and the 30th days, resulting in a total of 10 possible assignments. So, in the first three weeks, all participants are in phase A. The duration of phase A will thus be different for each subject. Phase A acts as a control and is therefore compared with phase B.
- Intervention phase (Phase B): Goal Management Training (Experimental): During the intervention phase (phase B), all included participants will have 6 sessions of Goal Management Training (GMT; twice per week) in which two individual chosen IADL-tasks will be subdivided into multiple steps under guidance of a therapist using the GMT method. In addition participants play the compensatory brain game in which they are challenged to apply the learned GMT strategy in an imaginary and safe environment.
  Interventions: Behavioral: Intervention during phase B: Compensatory brain game supporting Goal Management Training intervention
- Follow-up period (No Intervention): A follow-up period of three weeks takes place after phase B. During this follow-up period, patients receive no intervention.

INTERVENTIONS:
Behavioral: Intervention during phase B: Compensatory brain game supporting Goal Management Training intervention — The investigational treatment is only given during the intervention phase (phase B), and consists of six treatment sessions. In the treatment sessions, patients learn and apply the GMT algorithm. This means that the multiple steps of the GMT as well as the actual performance of the IADL-task goals will be learned under guidance of a therapist. In order to facilitate generalization, patients will learn to use the algorithm during the performance of untrained tasks by playing the treatment supporting Plan Game. Because of this, patients are able to practice the application of the GMT algorithm independently at their own home. Besides, the intervention also includes a Plan Tool. This is a mobile application that can be used as an aid during the performance of (instrumental) activities of daily living (IADL) tasks in order to perform activities more independently. The GMT treatment sessions are given twice a week (max. 60 minutes for each attendance).
  Arms: Intervention phase (Phase B): Goal Management Training

SUMMARY:
The main cognitive complaint in brain-injured patients is often the everyday disorganization caused by executive function (EF) deficits. In order to minimize the everyday disorganization, effective EF interventions are required. Interventions which incorporate compensatory strategies have the potential to enable patients to minimize disabilities, minimize participation problems and to function more independently in daily life. A well-known evidence-based intervention that incorporates compensatory strategies is Goal Management Training (GMT). GMT entails learning and applying an algorithm, in which a daily task is subdivided into multiple steps to handle executive difficulties of planning, and problem solving. To adopt the GMT strategy and ensure maximal profitability for patients, they have to learn to use the algorithm in different situations and tasks. Therefore, GMT is a comprehensive, time-consuming and thus labour-intensive treatment. Along with this, brain games become increasingly attractive as an (add-on) intervention, most notably in an effort to develop home-based personalized care. Until now, however, the rationale behind brain games is based on what can be considered the restorative approach (i.e. strengthening of executive problems) rather than practicing compensatory strategies, with little or no transfer to improvements in daily life functioning. This study therefore aims to assess the potential of a newly developed Brain Game, based on compensatory strategies, as an add-on to GMT to develop a shortened and partly home-based GMT intervention. The primary objective of this study is to assess whether the use of a compensatory brain game supported GMT treatment could be of interest in people with EF deficits after ABI, to improve goal achievement, their executive function performance during goal-related tasks, and their executive performance during an ecological valid shopping task. The study will be a multiple-baseline across individuals single-case experimental design (SCED). The study population consists of patients referred for outpatient cognitive rehabilitation. Participants eligible for the study must have executive deficits due to Acquired Brain Injury (ABI) of nonprogressive nature (i.e. TBI, stroke), with a minimum time post-onset of 3 months. Age has to be between 18 and 75 and participants have to live independently at home. Executive deficits will be assessed by extensive neuropsychological examination. Participants will be recruited from the outpatient clinic and the department of neurorehabilitation of Klimmendaal and Vogellanden. Four participants will be recruited.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 - 75 years
* Non-progressive acquired brain injury
* Minimal time post-onset of 3 months
* Outpatient rehabilitation
* Living independently at home
* Executive deficits (as determined on a neuropsychological assessment)

Exclusion Criteria:

* Inability to speak/understand the Dutch language
* Severe psychiatric problems (history)
* Neurodegenerative disorders
* Substance abuse
* Severe cognitive comorbidity (i.e. dementia)
* Aphasia
* Neglect
* No access to a smartphone, and laptop or tablet
* Unable to look at a computer screen for 15 minutes
* Unable to operate a keyboard or computer mouse

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2023-04-07 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in performance on the Oxford Multiple Errands Test- Dutch version (OxMET-NL) from phase A to phase B | The target behavior (i.e. performance on the OxMET-NL) will be measured repeatedly, two times a week, for the duration of phase A (3 to 5 weeks) and phase B (3 weeks)
  The target behavior will be assessed repeatedly, on a minimum of six occasions in phase A and B, in accordance with the recommendations of the What Works Clearinghouse and RoBiNT criteria (Tate et al., 2013). The OxMET-NL task is a computer-tablet based version of the Multiple Errands Test and is scored automatically. The task requires patients to buy six items and to answer two questions.

SECONDARY OUTCOMES:
Change on the Visual Analogue Scale (VAS) from phase A to phase B to follow-up | The VAS will be assessed repeatedly, two times a week, for the duration of phase A (3 to 5 weeks), phase B (3 weeks) and follow-up (3 weeks)
  Subjective experience of strategy use in daily life and during the performance of instrumental activities of daily living (IADL).
Change in performance on treatment goals as measured with the Goal Attainment Scale (GAS) | pre-intervention, immediately following intervention and at three weeks follow-up
  GAS is a mathematical technique for quantifying the achievement of goals set, used in rehabilitation. GAS is described as a method of scoring the extent to which patient's individual goals are achieved in the course of intervention. In effect, each patient has a own outcome measure, but this is scored in a standardized way as to allow statistical analysis. The achievement of each goal (IADL-task) can be measured on a 5-point scale ranging from -2 to +2. Outcomes can be quantified in a single aggregated goal attainment score. This method gives a numerical T-score which is normally distributed about a mean of 50 (if the goals are achieved precisely) with a standard deviation of around this mean of 10 (if the goals are overachieved or underachieved).
Change in performance on two trained IADL task (treatment goals) | pre-intervention, immediately following intervention and at three weeks follow-up
  Performance on two treatment goals is measured with a standardised scale which is similar to the one used by Bertens et al. (2015) and Dechamps et al. (2011). The tasks will be divided into multiple steps using the GMT method. Each task step will be assessed following a 3-point scale (ranging from 2=competent to 0=deficit). Total scores per task will be adjusted to a 100-point scale using the following formula: performance = (total score / (number of steps × 2)) × 100. Thus, a performance of 100% indicating perfect IADL task performance.
Change in everyday difficulties in activities/participation as measured on the Daily Living Questionnaire (DLQ-R-NL) | pre-intervention, immediately following intervention and at three weeks follow-up
  The Dutch version of the Daily Living Questionnaire measures how much mental or cognitive difficulty the participant generally has by performing daily activities.
Change in strategy use during the performance of trained and untrained IADL tasks | pre-intervention, immediately following intervention and at three weeks follow-up
  A self-designed questionnaire to examine self-reported strategy use will also be administered after the performance of the trained and untrained IADL tasks, based on the strategy questionnaire used by Frankenmolen, Fasotti, Kessels & Oosterman (2018), in order to measure strategy use in a traditional memory task. First, participants are openly asked which strategies they use during the performance of an IADL task. Subsequently, they are given a list with possible strategy components of GMT that one could use to perform a task and are asked to place a check mark next to each strategy that they had used.
Change in subjective experience of strategy use in daily life | pre-intervention, immediately following intervention and at three weeks follow-up
  GMT strategy use is assessed through an adjustment of the Strategy Use Inventory; SUI (Koning-Haanstra, Berg, & Deelman, 1990). Participants have to indicate how often they use a certain strategy in daily life situations using a 5-point rating scale ranging from 1 (never) to 5 (often). Average item scores are calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Elise Verhoog, MSc, Principal Investigator — Donders Centre for Cognitive Neuroimaging
Locations (1):
- Klimmendaal Revalidatiespecialisten, Arnhem, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided